CLINICAL TRIAL: NCT03580044
Title: A PROSPECTIVE, RANDOMIZED,OPEN-LABEL, COMPARATIVE STUDY TO ASSESS THE EFFICACY, SAFETY AND TOLERABILITY OF AZTREONAM- AVIBACTAM (ATM-AVI) AND BEST AVAILABLE THERAPY FOR THE TREATMENT OF SERIOUS INFECTIONS DUE TO MULTI-DRUG RESISTANT GRAM- NEGATIVE BACTERIA PRODUCING METALLO -Β-LACTAMASE (MBL)
Brief Title: Efficacy, Safety, and Tolerability of ATM-AVI in the Treatment of Serious Infection Due to MBL-producing Gram-negative Bacteria
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment of patients with serious infections caused by gram-negative bacteria producing MBL has been challenging. Date study terminated: 16-Dec-2022.
Sponsor: Pfizer (Industry)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C3601009; 2017-004544-38 (EudraCT Number); ASSEMBLE (Other: Alias Study Number)
Record Dates: First submitted 2018-06-04; First posted 2018-07-09 (Actual); Results first posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Serious Bacterial Infection
Keywords: Serious bacterial infection; cIAI; HAP/(VAP; cUTI; BSI; MBL

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ATM- AVI Aztreonam- Avibactam (ATM-AVI) Active Treatment Arm (Experimental)
  Interventions: Combination Product: ATM-AVI
- Best Available Therapy (BAT) Comparator Treatment Arm (Active Comparator)
  Interventions: Drug: BAT

INTERVENTIONS:
Combination Product: ATM-AVI — ATM-AVI doses (loading, extended loading and maintenance) and the dosing frequency of the maintenance dose are dependent on renal function. Subjects will be given a loading dose of 500 mg ATM plus 167 mg AVI or 675 mg ATM plus 225 mg AVI over a period of 30 minutes. This treatment will immediately be followed by an extended loading dose of 1500 mg ATM plus 500 mg AVI or 675 mg ATM plus 225 mg AVI over a period of 3 hours. Then there will be a 3 hour or 5 hour gap. Subjects will receive a maintenance dose of 1500 mg ATM plus 500 mg AVI every 6 hours or 750 mg ATM plus 250 mg AVI every 6 hours, or 675 mg ATM plus 225 mg AVI every 8 hours. Subjects with cIAI will also receive Metronidazole (MTZ) 500 mg IV q8h over 60 minutes. The first dose of MTZ will be started immediately after the extended loading dose of ATM-AVI has completed and treatment will be continued until the end of the treatment period.
  Other Names: Aztreonam- Avibactam
  Arms: ATM- AVI Aztreonam- Avibactam (ATM-AVI) Active Treatment Arm
Drug: BAT — The comparator treatment in this study is best available therapy (BAT) based upon site practice and local epidemiology. The choice of BAT (monotherapy or combination) for each subject must be recorded prior to randomization. If the chosen BAT does not provide adequate anaerobic coverage for cIAI subjects MTZ is to be administered as a co therapy. BAT dose, frequency, dose adjustments with renal impairment will be based on per local package inserts.
  Other Names: Best Available Therapy
  Arms: Best Available Therapy (BAT) Comparator Treatment Arm

SUMMARY:
Phase 3 study to determine the efficacy, safety, and tolerability of aztreonam- avibactam (ATM- AVI) versus best available therapy (BAT) in the treatment of hospitalized adults with complicated intra-abdominal infections (cIAI), nosocomial pneumonia (NP) including hospital acquired pneumonia (HAP) and ventilator associated pneumonia (VAP), complicated urinary tract infections (cUTI), or bloodstream infections (BSI) due to metallo-β-lactamase (MBL)- producing Gram-negative bacteria.

DETAILED DESCRIPTION:
This is a prospective, randomized, multicenter, open-label, parallel group, comparative study to determine the efficacy, safety, and tolerability of aztreonam- avibactam (ATM- AVI) versus best available therapy (BAT) in the treatment of hospitalized adults with complicated intra-abdominal infections (cIAI), nosocomial pneumonia (NP) including hospital acquired pneumonia (HAP) and ventilator associated pneumonia (VAP), complicated urinary tract infections (cUTI), or bloodstream infections (BSI) due to metallo-β-lactamase (MBL)- producing Gram-negative bacteria.

The study will randomize approximately 60 subjects in a 2:1 randomization scheme (ATM-AVI: BAT) with infections due to MBL-producing Gram-negative bacteria. Molecular testing at the central microbiology laboratory will be performed to confirm the MBL status of the organism upon study completion or at pre-designated intervals.

The study will consist of a Screening Visit (Visit 1), a Baseline visit (Visit 2) on Day 1 of the study treatment, ongoing treatment visits (Visits 3 to 15) from Day 2 to Day 14, an End of Treatment (EOT) visit (Visit 16) within 24 hours after the last infusion, a Test of Cure (TOC) visit (Visit 17) on Day 28 (±3 days) and a Late Follow Up (LFU) visit (Visit 18) on Day 45 (±3 days).

Subjects will be stratified at randomization based on infection type (cIAI, HAP/VAP, cUTI or BSI). The number of subjects with cUTI will be no more than approximately 75% of the study population.

After obtaining written informed consent and confirming eligibility, subjects will be randomized in a 2:1 ratio to the ATM AVI treatment arm or the BAT treatment arm according to a central randomization schedule (approximately 40 (ATM AVI) and approximately 20 (BAT) subjects per group).

The duration of treatment is 5 to 14 days for cIAI, cUTI and BSI and 7 to 14 days for HAP/VAP. Each subject is expected to complete the study, including the LFU visit. The precise duration of treatment will be determined by the investigator based on the subject's severity of infection and subsequent response to treatment.

For subjects randomized to ATM AVI treatment arm, sparse blood samples will be collected for population pharmacokinetic (PK) assessments and PK/pharmacodynamic (PD) relationships will be evaluated in subjects where plasma samples and microbiological response data have been collected.

ELIGIBILITY:
Inclusion Criteria All Subjects

1. Subject must be ≥18 years of age.
2. Evidence of a personally signed and dated informed consent document indicating that the subject or a legally acceptable representative has been informed of all pertinent aspects of the study.
3. Subjects must have a confirmed diagnosis of serious bacterial infection, specifically cIAI, HAP/VAP, cUTI, or BSI requiring administration of IV antibacterial therapy.
4. Subjects must have an MBL- positive Gram- negative bacteria (an Enterobacteriaceae and/or Stenotrophomonas maltophilia for which the imipenem or meropenem MIC is ≥ 4 µg/mL), that was isolated from an appropriate specimen obtained within 7 days prior to screening.
5. Female subject of childbearing potential must have a negative serum or urine pregnancy test, with sensitivity of at least 25 mIU/mL.
6. Subjects who have received more than 48 hours of an appropriate prior systemic antibiotic[s] for a carbapenem non -susceptible pathogen may be enrolled if they demonstrate worsening or lack of improvement of objective symptoms or signs of infection (Note: antibiotic[s] is considered appropriate if microbiological susceptibility test results show that all carbapenem non -susceptible pathogens are susceptible to the systemic antibiotic[s] received).

Additional Inclusion Criteria- cIAI Subjects

1. Subject must have a specimen obtained from an abdominal source during a surgical intervention within 7 days prior to screening from which a study qualifying pathogen was isolated upon culture. Surgical intervention includes open laparotomy, percutaneous drainage of an abscess, or laparoscopic surgery.
2. The subject has at least 1 of the following diagnosed during the surgical intervention:

   • Cholecystitis with gangrenous rupture or perforation or progression of the infection beyond the gallbladder wall;

   • Diverticular disease with perforation or abscess;
   * Appendiceal perforation or peri-appendiceal abscess;
   * Acute gastric or duodenal perforations, only if operated on >24 hours after diagnosis;
   * Traumatic perforation of the intestines, only if operated on >12 hours after diagnosis;
   * Other secondary peritonitis (not primary/ spontaneous bacterial peritonitis associated with cirrhosis or chronic ascites);
   * Intra abdominal abscess (including of the liver and spleen provided that there is extension beyond the organ with evidence of intra peritoneal involvement).
3. Subject has at least 1 of the following signs / symptoms from each of the following 2 groups:

   • Group A: Evidence of systemic inflammatory response:

   • Documented fever (defined as body temperature ≥38°C) or hypothermia (with a rectal core body temperature ≤35°C);

   • Elevated white blood cells (WBC) (>12000 cells/µL);

   • Systolic blood pressure (SBP) <90 mmHg or mean arterial pressure (MAP) <70 mmHg, or a SBP decrease of >40 mmHg;

   • Increased heart rate ( >90 beats per minute [bpm]) and respiratory rate (>20 breaths/min);

   • Hypoxemia (defined as oxygen [O2] saturation <95% by pulse oximetry);

   • Altered mental status.

   • Group B: Physical findings consistent with intra abdominal infection, such as:

   • Abdominal pain and/or tenderness, with or without rebound;

   • Localized or diffuse abdominal wall rigidity;

   • Abdominal mass.

Additional Inclusion Criteria - HAP/VAP Subjects

1. Onset of symptoms >48 hours after admission or <7 days after discharge from an inpatient care facility (for which the duration of admission was >3 days).
2. New or worsening infiltrate on chest X- ray (or computerized tomography [CT]- scan) obtained within 48 hours prior to randomization.
3. At least 1 of the following:

   * Documented fever (temperature ≥38°C) or hypothermia (rectal/core temperature ≤35°C);
   * WBC ≥10,000 cells/mm3, leukopenia with total WBC ≤4500 cells/mm3, or >15% immature neutrophils (bands) noted on peripheral blood smear.
4. At least 2 of the following:

   • A new cough (or worsening of cough at Baseline);

   • Production of purulent sputum or purulent endotracheal secretions;

   • Auscultatory finding consistent with pneumonia/pulmonary consolidation (eg, rales, rhonchi, bronchial breath sounds, dullness on percussion, egophony);

   • Dyspnea, tachypnea, or hypoxemia (O2 saturation <90% or partial pressure of O2 [pO2]<60 mmHg while breathing room air);

   • Need for acute changes in the ventilator support status/system to enhance oxygenation, as determined by worsening oxygenation (arterial blood gas [ABG] or pO2 in arterial blood [PaO2]/fraction of inspired O2 [FiO2]) or needed changes in the amount of positive end expiratory pressure.
5. Subjects must have a respiratory specimen obtained within 7 days prior to screening for Gram stain and culture from which a study qualifying pathogen was isolated upon culture. This includes culture of either an expectorated sputum or a specimen of respiratory secretions obtained by endotracheal aspiration in intubated subjects, or by bronchoscopy with bronchoalveolar lavage (BAL), mini BAL or protected specimen brush (PSB) sampling.

Additional Inclusion Criteria - cUTI Subjects

1. Subject had urine within 7 days prior to screening that cultured positive; containing ≥10^5 colony forming unit (CFU)/mL of at least 1 carbapenem non susceptible, MBL positive Gram-negative bacteria, ie, the isolate from the study qualifying culture.
2. Subject had pyuria in the 7 days prior to screening as determined by a midstream clean catch or catheterized urine specimen with ≥10 white blood cells (WBCs) per HighPower Field (HPF) on standard examination of urine sediment or ≥10 WBCs/mm3 in unspun urine.
3. Subject demonstrates either acute pyelonephritis or complicated lower UTI without pyelonephritis as defined by the following criteria:

   a. Acute pyelonephritis indicated by flank pain (which must have onset or worsened within 7 days of enrollment) or costovertebral angle tenderness on examination and at least 1 of the following: i) Fever, defined as body temperature ≥38°C (with or without patient symptoms of rigor, chills, or warmth); ii) Nausea and/or vomiting. OR b. Complicated lower UTI, as indicated by qualifying symptoms plus at least 1 complicating factor as follows: i) Qualifying symptoms: subject must have at least 2 of the following symptoms with at least 1 symptom from Group A:

   • Group A symptoms include dysuria, urgency, frequency, and or suprapubic pain;

   • Group B symptoms include fever (defined as body temperature ≥38°C with or without patient symptoms of rigor, chills, warmth), nausea, and/or vomiting.

   ii) Complicating factors: subject must have at least 1 of the following complicating factors:

   • Documented history of urinary retention (male subjects);

   • Obstructive uropathy that is scheduled to be medically or surgically relieved during study therapy and before the EOT;

   • Functional or anatomical abnormality of the urogenital tract, including anatomic malformations or neurogenic bladder, or with a postvoid residual urine volume of at least 100 mL;

   • Use of intermittent bladder catheterization or presence of an indwelling bladder catheter for at least 48 hours;

   • Urogenital procedure (such as cystoscopy or urogenital surgery) within the 7 days prior to obtainment of the specimen used for the study qualifying culture.

   Additional Inclusion Criteria - BSI Subjects

<!-- -->

1. Subject has a confirmed diagnosis of primary BSI or catheter related BSI (CR- BSI).
2. Signs and symptoms of systemic infection characterized by at least one of the following:

   1. Chills, rigors, or fever (temperature of ≥38.0°C or ≥100.4°F);
   2. Elevated white blood cell count (≥10,000/mm3) or left shift (>15% immature polymorphonuclear leukocytes (PMNs)).

Exclusion Criteria All Subjects

1. History of serious allergic reaction (anaphylaxis, angioedema, bronchospasm, hypersensitivity) to any systemic antibacterial allowed per protocol.
2. Subject has a concurrent infection that may interfere with the evaluation of response to the study antibiotics.
3. Subject has a need for effective concomitant systemic antibacterials in addition to those allowed per protocol for the diagnoses under study.
4. Estimated CrCL ≤15 mL/min or anticipated requirement for dialysis during the study.

Additional Exclusion Criteria - cIAI Subjects

1. Subject has infections limited to the hollow viscous, such as simple cholecystitis, gangrenous cholecystitis without rupture, and simple appendicitis, or has acute suppurative cholangitis, infected necrotizing pancreatitis, or pancreatic abscess.
2. Subject has abdominal wall abscess or small bowel obstruction without perforation or ischemic bowel without perforation.
3. Subject has a cIAI managed by staged abdominal repair (STAR), or "open abdomen" technique, or marsupialization. This criterion is intended to exclude subjects in whom the abdomen is left open, particularly those for whom re operation is planned.

Additional exclusion criteria - cUTI Subjects 1. Subjects with suspected or confirmed complete obstruction of any portion of the urinary tract, perinephric or intrarenal abscess, or prostatitis, or history of any illness that, in the opinion of the investigator, may confound the results of the study or pose additional risk in administering the study therapy to the subject.

2. Any recent history of trauma to the pelvis or urinary tract.

Additional exclusion criteria - BSI Subjects

1. Subject has a prosthetic cardiac valve or synthetic endovascular graft. 2. Subject has a suspected or documented medical condition with well-defined requirement for prolonged antibiotic treatment (eg, infectious endocarditis, osteomyelitis/septic arthritis, undrainable/undrained abscess, unremoveable/unremoved prosthetic associated infection).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-12-25 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (42):
- Banner University Medical Center Tucson, Tucson, Arizona, United States
- Hospital San Roque, Córdoba, Argentina
- China (6):
  - The First Affiliated Hospital of Shantou University Medical College, Shantou, Guangdong
  - Hunan Province People's Hospital, Changsha, Hunan
  - Baotou Central Hospital, Baotou, Inner Mongolia
  - Huashan Hospital Fudan University, Shanghai, Shanghai Municipality
  - The First Hospital of Kunming, Kunming, Yunnan
  - The First Hospital of Kunming, Kunming
- Greece (6):
  - General Hospital of Athens "Evangelismos", Athens
  - General and Chest Diseases Hospital "Sotiria", Athens
  - General Hospital of Athens "Laiko",, Athens
  - University General Hospital "ATTIKON", Medicine and Infectious Diseases, Athens
  - University General Hospital of Heraklion, Heraklion, Crete
  - University General Hospital of Larissa, Larissa
- India (5):
  - Government medical College, Kozhikode, Kerala
  - Deenanath Mangeshkar Hospital And Research Centre, Pune, Maharashtra
  - S.R.Kalla Memorial Gastro & General Hospital, Jaipur, Rajasthan
  - Apollo Hospitals Enterprise Limited, Chennai, Tamil Nadu
  - Victoria Hospital, Bangalore Medical College and Research Institute, Bangalore
- Malaysia (2):
  - Hospital Kuala Lumpur, Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
- Hospital Civil de Guadalajara "Fray Antonio Alcalde", Guadalajara, Jalisco, Mexico
- Philippines (4):
  - Davao Doctors Hospital, Davao City
  - Makati Medical Center, Makati City
  - Manila Doctors Hospital, Manila
  - St. Luke's Medical Center, Quezon City
- Romania (5):
  - Institutul National de Boli Infectioase "Prof. Dr. Matei Bals", Bucharest
  - Spitalul Clinic de Boli Infectioase si Tropicale "Dr. Victor Babes", Bucharest
  - Spitalul Clinic de Boli Infectioase Cluj Napoca, Cluj-Napoca
  - Spitalul Clinic de Boli Infectioase "Sf. Parascheva" Iasi, Iași
  - Spitalul Clinic Judetean de Urgenta "Pius Brinzeu", Timișoara
- Russia (4):
  - SBHI of the city of Moscow "N.I.Pirogov City Clinical Hospital # 1", Moscow
  - OGBUZ "Smolensk Regional Clinical Hospital", Smolensk
  - FSBEI of HE "Smolensk State Medical University" of the Ministry of Health of the RF, Smolensk
  - SRI of Antimicrobial Chemotherapy, Smolensk
- Taiwan (3):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
- Thailand (4):
  - Faculty of Medicine Siriraj Hospital, Bangkoknoi, Bangkok
  - Bamrasnaradura Infectious Disease Institute (BIDI), Muang, Changwat Nonthaburi
  - Songklanagarind Hospital, Prince of Songkla University, Hat Yai, Changwat Songkhla
  - Srinagarind Hospital, Division of lnfectious Disease and Tropical Medicine, Muang, Khonkaen

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Raber SR, Xie R, Rogers H, Soto E, Arhin FF, Stone GG, Leister-Tebbe H, Chow JW. Microbiological, Clinical, and Pharmacokinetic/Pharmacodynamic Data to Support EUCAST Aztreonam-Avibactam Minimum Inhibitory Concentration Susceptibility Breakpoints Against Enterobacterales. Infect Dis Ther. 2026 Jan;15(1):183-195. doi: 10.1007/s40121-025-01267-3. Epub 2025 Nov 21. PMID 41269522
- [Derived] Xie R, Rogers H, Chow JW, Soto E, Raber SR. Population pharmacokinetic/pharmacodynamic modeling to optimize aztreonam-avibactam dose regimens for adult patients. Antimicrob Agents Chemother. 2025 Aug 6;69(8):e0195024. doi: 10.1128/aac.01950-24. Epub 2025 Jun 18. PMID 40530972
- [Derived] Das S, Riccobene T, Carrothers TJ, Wright JG, MacPherson M, Cristinacce A, McFadyen L, Xie R, Luckey A, Raber S. Dose selection for aztreonam-avibactam, including adjustments for renal impairment, for Phase IIa and Phase III evaluation. Eur J Clin Pharmacol. 2024 Apr;80(4):529-543. doi: 10.1007/s00228-023-03609-x. Epub 2024 Jan 22. PMID 38252170
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3601009

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who were hospitalized with a diagnosis of complicated intra-abdominal infection (cIAI), nosocomial pneumonia (NP) including hospital-acquired pneumonia (HAP) and ventilator-associated pneumonia (VAP), complicated urinary tract infection (cUTI), or bloodstream infections (BSI) due to Metallo-beta-Lactamase (MBL)- producing Gram-negative bacteria were enrolled. This study was conducted across 9 countries from 25 Dec-2020 to 23-Jan-2023.
Pre-assignment Details: A total of 15 participants signed the informed consent form and were randomized in the study. The study was terminated as recruitment of participants with serious infections caused by gram-negative bacteria producing MBL was challenging.
Groups:
- Aztreonam- Avibactam (ATM- AVI): Participants were administered a loading dose of aztreonam- avibactam (ATM-AVI) by intravenous (IV) infusion over 30 minutes immediately followed by an extended loading dose of ATM-AVI by infusion over 3 hours, and then started a maintenance dose of ATM-AVI by IV infusion over 3 hours on Day 1. Participants with creatinine clearance >50 milliliters per minute (mL/min) and >30 to 50 mL per minute were administered maintenance dose once every 6 hours for maximum of 14 days. Participants with creatinine clearance >15 to 30 mL/min were administered maintenance dose once every 8 hours for maximum of 14 days. Participants with cIAI also received metronidazole (MTZ) 500 milligram (mg) every 8 hours by IV infusion over 60 minutes.
- Best Available Therapy (BAT): Participants who were hospitalized with a diagnosis of cIAI, NP, HAP, VAP, cUTI or BSI received Best Available Therapy (BAT) based upon site practice and local epidemiology for a maximum of 14 days. Participants with cIAI in the BAT arm received metronidazole if BAT did not provide adequate anaerobic coverage.
Period: Overall Study
Arm/Group | Aztreonam- Avibactam (ATM- AVI) | Best Available Therapy (BAT)
Started | 12 | 3
Treated | 12 | 2
Completed | 9 | 1
Not Completed | 3 | 2
Not completed — Death | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) analysis set included all randomized participants regardless of receipt of study drug. Participants were analyzed according to the treatment to which they were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Aztreonam- Avibactam (ATM- AVI) | Best Available Therapy (BAT) | Total
Number analyzed (Participants) | 12 | 3 | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.6 (17.14) | 65.7 (6.66) | 58.4 (15.85)
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 8 | 2 | 10
  65-74 years | 3 | 1 | 4
  75-84 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 8 | 1 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 11 | 3 | 14
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 6 | 1 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 2 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Cure at the Test of Cure (TOC) Visit -Microbiological Intent to Treat (Micro-ITT) Analysis Set
Description: Clinical cure was defined as improvement in baseline signs and symptoms such that no further antimicrobial treatment was required for the index infection (i.e., cIAI, cUTI, HAP/VAP or BSI) after study treatment. Also for cIAI participants, no unplanned drainage or surgical intervention was necessary since the initial procedure. The clinical response assessment was determined by a blinded independent adjudication committee. 95% confidence interval (CI) was calculated using Jeffrey's method.
Time Frame: Day 28
Population: Micro-ITT analysis set was a subset of the ITT analysis set and included all participants who had at least 1 MBL-positive Gram-negative baseline pathogen from an adequate specimen at the start of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Aztreonam- Avibactam (ATM- AVI) | Best Available Therapy (BAT)
Number analyzed (Participants) | 12 | 3
Percentage of participants | 41.7 [18.0 to 68.8] | 0.0 [NA to NA] — 95% CI could not be calculated due to insufficient number of participants with events.

2. Secondary Outcome: Percentage of Participants With Clinical Cure at the TOC Visit-Microbiologically Evaluable (ME) Analysis Set
Description: Clinical cure was defined as improvement in baseline signs and symptoms such that no further antimicrobial treatment was required for the index infection (i.e., cIAI, cUTI, HAP/VAP or BSI) after study treatment. Also, for cIAI participants, no unplanned drainage or surgical intervention was necessary since the initial procedure. The clinical response assessment was determined by a blinded independent adjudication committee. 95% CI was calculated using Jeffrey's method.
Time Frame: Day 28
Population: ME analysis set: Participants from micro-ITT who received at least 48 hours of study therapy or <48 hours before discontinuation due to an adverse event, no concomitant antibiotics against baseline MBL positive pathogens between first dose of study therapy and TOC (excluding participants with failed study therapy requiring additional antibiotics), had baseline organisms confirmed by central microbiological testing (except when locally confirmed) and no indeterminate clinical outcomes at TOC.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Aztreonam- Avibactam (ATM- AVI) | Best Available Therapy (BAT)
Number analyzed (Participants) | 9 | 1
Percentage of participants | 55.6 [25.4 to 82.7] | 0.0 [NA to NA] — 95% CI could not be calculated due to insufficient number of participants with events.

3. Secondary Outcome: Percentage of Participants With Clinical Cure at the End of Treatment (EOT) Visit- Micro-ITT Analysis Set
Description: Clinical cure was defined as improvement in baseline signs and symptoms such that no further antimicrobial treatment was required for the index infection (i.e., cIAI, cUTI, HAP/VAP or BSI) after study treatment. Also for cIAI participants, no unplanned drainage or surgical intervention was necessary since the initial procedure. The clinical response assessment was determined by a blinded independent adjudication committee. 95% CI was calculated using Jeffrey's method.
Time Frame: Up to 24 hours after the last infusion on Day 14
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Aztreonam- Avibactam (ATM- AVI) | Best Available Therapy (BAT)
Number analyzed (Participants) | 12 | 3
Percentage of participants | 58.3 [31.2 to 82.0] | 0.0 [NA to NA] — 95% CI could not be calculated due to insufficient number of participants with events.

4. Secondary Outcome: Percentage of Participants With Clinical Cure at the EOT Visit- ME Analysis Set
Description: as for outcome 3
Time Frame: Up to 24 hours after the last infusion on Day 14
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Aztreonam- Avibactam (ATM- AVI) | Best Available Therapy (BAT)
Number analyzed (Participants) | 9 | 1
Percentage of participants | 66.7 [34.8 to 89.6] | 0.0 [NA to NA] — 95% CI could not be calculated due to insufficient number of participants with events.

5. Secondary Outcome: Percentage of Participants With a Favorable Per Participant Microbiological Response at EOT Visit-Micro-ITT Analysis Set
Description: Favorable microbiological response was defined as eradication or presumed eradication. Eradication was defined as absence (or urine quantification <10^3 colony forming units per milliliter [CFU/mL] for cUTI participants) of causative pathogen from an appropriately obtained specimen at the site of infection. Presumed eradication was defined as repeat culture of specimens were not performed/clinically indicated in a participant who had a clinical response of cure (specific to cIAI and HAP/VAP participants).
Time Frame: Up to 24 hours after the last infusion on Day 14
Population: Micro-ITT analysis set was a subset of the ITT analysis set and included all participants who had at least 1 MBL-positive Gram-negative baseline pathogen from an adequate specimen at the start of study treatment. Participants with a per participant response of Indeterminate were excluded from this analysis. Here 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Aztreonam- Avibactam (ATM- AVI) | Best Available Therapy (BAT)
Number analyzed (Participants) | 11 | 1
Percentage of participants | 81.82 | 0.0

6. Secondary Outcome: Percentage of Participants With a Favorable Per Participant Microbiological Response at TOC Visit-Micro-ITT Analysis Set
Description: as for outcome 5
Time Frame: Day 28
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | Aztreonam- Avibactam (ATM- AVI) | Best Available Therapy (BAT)
Number analyzed (Participants) | 10 | 1
Percentage of participants | 60.00 | 0.0

7. Secondary Outcome: Percentage of Participants With a Favorable Per Participant Microbiological Response at EOT Visit-ME Analysis Set
Description: Favorable microbiological response was defined as eradication or presumed eradication. Eradication was defined as absence (or urine quantification <10^3 CFU/mL for cUTI participants) of causative pathogen from an appropriately obtained specimen at the site of infection. Presumed eradication was defined as repeat culture of specimens were not performed/clinically indicated in a participant who had a clinical response of cure (specific to cIAI and HAP/VAP participants).
Time Frame: Up to 24 hours after the last infusion on Day 14
Population: ME analysis set: Participants from micro-ITT who received at least 48 hours of study therapy or <48 hours before discontinuation due to an adverse event; no concomitant antibiotics against baseline MBL positive pathogens between first dose of study therapy and TOC (excluding participants with failed study therapy requiring additional antibiotics), had baseline organisms confirmed by central microbiological testing (except when locally confirmed) and no indeterminate clinical outcomes at TOC.
Measure: Number; unit: Percentage of participants
Arm/Group | Aztreonam- Avibactam (ATM- AVI) | Best Available Therapy (BAT)
Number analyzed (Participants) | 9 | 1
Percentage of participants | 66.67 | 0.00

8. Secondary Outcome: Percentage of Participants With a Favorable Per Participant Microbiological Response at TOC Visit-ME Analysis Set
Description: as for outcome 7
Time Frame: Day 28
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Aztreonam- Avibactam (ATM- AVI) | Best Available Therapy (BAT)
Number analyzed (Participants) | 9 | 1
Percentage of participants | 66.7 | 0.00

9. Secondary Outcome: Percentage of Pathogens According to Favourable Per-Pathogen Microbiological Response at the EOT Visit-Micro-ITT Analysis Set
Description: as for outcome 7
Time Frame: Up to 24 hours after the last infusion on Day 14
Population: Micro-ITT analysis set was a subset of the ITT analysis set and included all participants who had at least 1 MBL-positive Gram-negative baseline pathogen from an adequate specimen at the start of study treatment. All pathogens reported under 'Overall Number of Pathogens Analyzed' contributed data to the table; however, may not have evaluable data for every row. Here, 'Number Analyzed (n)'= pathogens evaluable for specified rows.
Measure: Number; unit: Percentage of pathogens
Units Other Than Participants: Pathogens
Arm/Group | Aztreonam- Avibactam (ATM- AVI) | Best Available Therapy (BAT)
Number analyzed (Participants) | 12 | 3
Number analyzed (Pathogens) | 18 | 3
Percentage of pathogens
  Enterobacterales: number analyzed (Pathogens) | 12 | 3
  Enterobacterales | 75.0 | 0.0
  Pseudomonas aeruginosa: number analyzed (Pathogens) | 2 | 0
  Pseudomonas aeruginosa | 50.0 |
  Stenotrophomonas maltophilia: number analyzed (Pathogens) | 3 | 0
  Stenotrophomonas maltophilia | 66.7 |
  Enterococcus faecium: number analyzed (Pathogens) | 1 | 0
  Enterococcus faecium | 100.0 |

10. Secondary Outcome: Percentage of Pathogens According to Favourable Per-Pathogen Microbiological Response at the TOC Visit-Micro-ITT Analysis Set
Description: as for outcome 7
Time Frame: Day 28
Population: Micro-ITT analysis set was a subset of the ITT analysis set and included all participants who had at least 1 MBL-positive Gram-negative baseline pathogen from an adequate specimen at the start of study treatment. All pathogens reported under 'Overall Number of Pathogens Analyzed' contributed data to the table; however, may not have evaluable data for every row. n= pathogens evaluable for specified rows.
Measure: Number; unit: Percentage of pathogens
Units Other Than Participants: Pathogens
Arm/Group | Aztreonam- Avibactam (ATM- AVI) | Best Available Therapy (BAT)
Number analyzed (Participants) | 12 | 3
Number analyzed (Pathogens) | 18 | 3
Percentage of pathogens
  Enterobacterales: number analyzed (Pathogens) | 12 | 3
  Enterobacterales | 50.0 | 0.00
  Pseudomonas aeruginosa: number analyzed (Pathogens) | 2 | 0
  Pseudomonas aeruginosa | 0.0 |
  Stenotrophomonas maltophilia: number analyzed (Pathogens) | 3 | 0
  Stenotrophomonas maltophilia | 33.3 |
  Enterococcus faecium: number analyzed (Pathogens) | 1 | 0
  Enterococcus faecium | 0.0 |

11. Secondary Outcome: Percentage of Pathogens According to Favourable Per-Pathogen Microbiological Response at the EOT Visit-ME Analysis Set
Description: Favorable microbiological response was defined as eradication or presumed eradication. Eradication was defined as absence (or urine quantification <10^3 CFU/mL for cUTI participants) of causative pathogen from an appropriately obtained specimen at the site of infection. Presumed eradication was defined as repeat culture of specimens were not performed/clinically indicated in a participant who had a clinical response of cure (specific to cIAI and HAP/VAP participants). ME analysis set comprised of participants from micro-ITT who received at least 48 hours or <48 hours of study therapy before discontinuation due to AE, no concomitant antibiotics against baseline MBL positive pathogens between 1st dose and TOC (excluding those with failed study therapy requiring additional antibiotics), had baseline organisms confirmed by central microbiological testing (except when locally confirmed); no indeterminate clinical outcomes at TOC.
Time Frame: Up to 24 hours after the last infusion on Day 14
Population: ME analysis set. All pathogens reported under 'Overall Number of Pathogens Analyzed' contributed data to the table; however, may not have evaluable data for every row. n= pathogens evaluable for specified rows.
Measure: Number; unit: Percentage of pathogens
Units Other Than Participants: Pathogens
Arm/Group | Aztreonam- Avibactam (ATM- AVI) | Best Available Therapy (BAT)
Number analyzed (Participants) | 9 | 1
Number analyzed (Pathogens) | 13 | 1
Percentage of pathogens
  Enterobacterales: number analyzed (Pathogens) | 10 | 1
  Enterobacterales | 80.0 | 0.0
  Stenotrophomonas maltophilia: number analyzed (Pathogens) | 2 | 0
  Stenotrophomonas maltophilia | 100.0 |
  Enterococcus faecium: number analyzed (Pathogens) | 1 | 0
  Enterococcus faecium | 100.0 |

12. Secondary Outcome: Percentage of Pathogens According to Favourable Per-Pathogen Microbiological Response at the TOC Visit-ME Analysis Set
Description: as for outcome 11
Time Frame: Day 28
Population: as for outcome 11
Measure: Number; unit: Percentage of pathogens
Units Other Than Participants: pathogens
Arm/Group | Aztreonam- Avibactam (ATM- AVI) | Best Available Therapy (BAT)
Number analyzed (Participants) | 9 | 1
Number analyzed (pathogens) | 13 | 1
Percentage of pathogens
  Enterobacterales: number analyzed (pathogens) | 10 | 1
  Enterobacterales | 60.0 | 0.0
  Stenotrophomonas maltophilia: number analyzed (pathogens) | 2 | 0
  Stenotrophomonas maltophilia | 50.0 |
  Enterococcus faecium: number analyzed (pathogens) | 1 | 0
  Enterococcus faecium | 0.0 |

13. Secondary Outcome: Percentage of Participants Who Died Within 28 Days From Randomization-ITT Analysis Set
Description: Percentage of participants who died due to any cause on or before 28 days after randomization were reported in this outcome measure.
Time Frame: From randomization up to Day 28
Population: ITT analysis set included all randomized participants regardless of receipt of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Aztreonam- Avibactam (ATM- AVI) | Best Available Therapy (BAT)
Number analyzed (Participants) | 12 | 3
Percentage of participants | 8.3 | 33.3

14. Secondary Outcome: Percentage of Participants Who Died Within 28 Days From Randomization- Micro ITT Analysis Set
Description: as for outcome 13
Time Frame: From randomization up to Day 28
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Aztreonam- Avibactam (ATM- AVI) | Best Available Therapy (BAT)
Number analyzed (Participants) | 12 | 3
Percentage of participants | 8.3 | 33.3

15. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events and Serious Adverse Events
Description: An adverse event (AE) was any untoward medical occurrence in a study participant administered a product or medical device; the event need not necessarily have a causal relationship with the treatment or usage. A serious adverse event (SAE) was any untoward medical occurrence at any dose that: resulted in death; was life-threatening (immediate risk of death); required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/ incapacity; resulted in congenital anomaly/birth defect; considered an important medical event. Treatment-emergent adverse event (TEAE) was any AE that started after the study medication start date and time.
Time Frame: From first dose of study treatment (Day 1) until late follow-up visit (Up to Day 45)
Population: Safety analysis set included all participants who received any amount of study treatment. Participants were analyzed according to the treatment they received.
Measure: Count of Participants; unit: Participants
Arm/Group | Aztreonam- Avibactam (ATM- AVI) | Best Available Therapy (BAT)
Number analyzed (Participants) | 12 | 2
Participants
  TEAEs | 11 | 2
  SAEs | 5 | 2

16. Secondary Outcome: Number of Participants With Vital Sign Abnormalities
Description: Vital signs included blood pressure and heart rate and were measured in a supine position after at least 10 minutes of rest for the participants. Criteria for vital sign abnormalities included: systolic blood pressure (SBP): value >150 millimeters of mercury (mmHg) and increase from baseline >=30 mmHg and value <90 and decrease from baseline ≥30. Diastolic BP (mm Hg) Value >100 and increase from baseline >= 20 and Value <50 and decrease from baseline >=20. Heart Rate (beats per minute [BPM]): Value <40 or >120.
Time Frame: From first dose of study treatment (Day 1) until TOC (Up to Day 28)
Population: Safety analysis set included all participants who received any amount of study treatment. Participants were analyzed according to the treatment they received. Here 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Aztreonam- Avibactam (ATM- AVI) | Best Available Therapy (BAT)
Number analyzed (Participants) | 11 | 2
Participants
  SBP: Value >150 and increase from baseline >=30 | 3 | 0
  SBP: Value <90 and decrease from baseline >=30 | 0 | 1
  DBP: Value >100 and increase from baseline >=20 | 0 | 0
  DBP: Value <50 and decrease from baseline >=20 | 0 | 0
  Heart Rate (BPM): <40 or >120 | 6 | 2

17. Secondary Outcome: Number of Participants With Abnormal Physical Examination Findings
Description: Physical examination included assessment of the following: abdomen, cardiovascular, ears, eyes, general appearance, head, lungs, lymph nodes, musculoskeletal, neurological, nose, skin and throat. Number of participants with abnormal physical examination findings for each body system is reported in this outcome measure.
Time Frame: Baseline (last non-missing value observed before start of treatment on Day 1), EOT (Up to 24 hours after the last infusion on Day 14), TOC (Day 28)
Population: Safety analysis set included all participants who received any amount of study treatment. Participants were analyzed according to the treatment they received. Here, 'Number Analyzed'= participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Aztreonam- Avibactam (ATM- AVI) | Best Available Therapy (BAT)
Number analyzed (Participants) | 12 | 2
Participants
  Abdomen - Baseline | 3 | 0
  Abdomen - End of Treatment: number analyzed (Participants) | 11 | 1
  Abdomen - End of Treatment | 4 | 0
  Abdomen -Test of cure: number analyzed (Participants) | 8 | 1
  Abdomen -Test of cure | 2 | 0
  Cardiovascular - Baseline | 1 | 2
  Cardiovascular - End of Treatment: number analyzed (Participants) | 11 | 1
  Cardiovascular - End of Treatment | 1 | 1
  Cardiovascular -Test of cure: number analyzed (Participants) | 8 | 1
  Cardiovascular -Test of cure | 0 | 1
  Ears- Baseline | 0 | 0
  Ears - End of Treatment: number analyzed (Participants) | 11 | 1
  Ears - End of Treatment | 0 | 0
  Ears-Test of cure: number analyzed (Participants) | 8 | 1
  Ears-Test of cure | 0 | 0
  Eyes - Baseline | 2 | 0
  Eyes - End of Treatment: number analyzed (Participants) | 11 | 1
  Eyes - End of Treatment | 3 | 0
  Eyes -Test of cure: number analyzed (Participants) | 8 | 1
  Eyes -Test of cure | 1 | 0
  General Appearance- Baseline | 5 | 1
  General Appearance - End of Treatment: number analyzed (Participants) | 11 | 1
  General Appearance - End of Treatment | 3 | 0
  General Appearance-Test of cure: number analyzed (Participants) | 8 | 1
  General Appearance-Test of cure | 0 | 0
  Head- Baseline | 2 | 0
  Head- End of Treatment: number analyzed (Participants) | 11 | 1
  Head- End of Treatment | 2 | 0
  Head- Test of cure: number analyzed (Participants) | 8 | 1
  Head- Test of cure | 0 | 0
  Lungs- Baseline | 4 | 1
  Lungs-End of Treatment: number analyzed (Participants) | 11 | 1
  Lungs-End of Treatment | 2 | 0
  Lungs-Test of cure: number analyzed (Participants) | 8 | 1
  Lungs-Test of cure | 1 | 0
  Lymph Nodes-Baseline | 0 | 0
  Lymph Nodes-End of Treatment: number analyzed (Participants) | 11 | 1
  Lymph Nodes-End of Treatment | 0 | 0
  Lymph Nodes-Test of cure: number analyzed (Participants) | 8 | 1
  Lymph Nodes-Test of cure | 0 | 0
  Musculoskeletal-Baseline | 3 | 2
  Musculoskeletal-End of Treatment: number analyzed (Participants) | 11 | 1
  Musculoskeletal-End of Treatment | 1 | 1
  Musculoskeletal-Test of cure: number analyzed (Participants) | 8 | 1
  Musculoskeletal-Test of cure | 1 | 1
  Neurological-Baseline | 8 | 1
  Neurological-End of Treatment: number analyzed (Participants) | 11 | 1
  Neurological-End of Treatment | 5 | 0
  Neurological-Test of cure: number analyzed (Participants) | 8 | 1
  Neurological-Test of cure | 3 | 0
  Nose-Baseline | 1 | 0
  Nose-End of Treatment: number analyzed (Participants) | 11 | 1
  Nose-End of Treatment | 0 | 0
  Nose-Test of cure: number analyzed (Participants) | 8 | 1
  Nose-Test of cure | 0 | 0
  Skin-Baseline | 5 | 0
  Skin-End of Treatment: number analyzed (Participants) | 11 | 1
  Skin-End of Treatment | 3 | 0
  Skin-Test of cure: number analyzed (Participants) | 8 | 1
  Skin-Test of cure | 1 | 0
  Throat-Baseline: number analyzed (Participants) | 11 | 2
  Throat-Baseline | 0 | 1
  Throat-End of Treatment: number analyzed (Participants) | 11 | 1
  Throat-End of Treatment | 1 | 0
  Throat-Test of cure: number analyzed (Participants) | 8 | 1
  Throat-Test of cure | 1 | 0

18. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Hematology Assessments
Description: Potential clinically significant criteria included: Hematocrit <0.7*lower limit of normal (LLN) and >30% Decrease from Baseline or >1.3*upper limit of normal (ULN) and >30% Increase from Baseline; Hemoglobin: <0.7*LLN and >30% Decrease from Baseline and>1.3*ULN and >30% Increase from Baseline;;Erythrocytes: <0.7*LLN and >30% Decrease from Baseline or >1.3*ULN and >30% Increase from Baseline; Leukocytes: <0.65*LLN and >60% Decrease from Baseline or >1.5*ULN and >100% Increase from Baseline; Basophils/Leukocytes, Eosinophils/Leukocytes and Monocytes/Leukocytes: >4.0*ULN and>300% Increase from Baseline; Lymphocytes/Leukocytes <0.25*LLN and >75% Decrease from Baseline and >1.5* ULN and >100% Increase from Baseline; Neutrophils/Leukocytes: <0.65*LLN and >75% Decrease from Baseline or >1.6*ULN and >100% Increase from Baseline; Platelets<0.65*LLN and >50% Decrease from Baseline or >1.5*ULN and >100% Increase from Baseline.
Time Frame: From first dose of study treatment (Day 1) until TOC (Up to Day 28)
Population: Safety analysis set included all participants who received any amount of study treatment. Participants were analyzed according to the treatment they received. All participants reported under 'Overall Number of Participants Analyzed' contributed data to the table but may not have evaluable data for every row. Here, 'Number Analyzed'= participants evaluable for specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Aztreonam- Avibactam (ATM- AVI) | Best Available Therapy (BAT)
Number analyzed (Participants) | 12 | 2
Participants
  Hematocrit: <0.7* LLN and >30% Decrease from Baseline: number analyzed (Participants) | 11 | 1
  Hematocrit: <0.7* LLN and >30% Decrease from Baseline | 0 | 0
  Hematocrit: >1.3* ULN and >30% Increase from Baseline: number analyzed (Participants) | 11 | 1
  Hematocrit: >1.3* ULN and >30% Increase from Baseline | 0 | 0
  Hemoglobin: <0.7* LLN and >30% Decrease from Baseline: number analyzed (Participants) | 11 | 1
  Hemoglobin: <0.7* LLN and >30% Decrease from Baseline | 0 | 0
  Hemoglobin: >1.3* ULN and >30% Increase from Baseline: number analyzed (Participants) | 11 | 1
  Hemoglobin: >1.3* ULN and >30% Increase from Baseline | 0 | 0
  Erythrocytes: <0.7* LLN and >30% Decrease from Baseline: number analyzed (Participants) | 11 | 1
  Erythrocytes: <0.7* LLN and >30% Decrease from Baseline | 0 | 0
  Erythrocytes: >1.3* ULN and >30% Increase from Baseline: number analyzed (Participants) | 11 | 1
  Erythrocytes: >1.3* ULN and >30% Increase from Baseline | 0 | 0
  Leukocytes: <0.65* LLN and >60% Decrease from Baseline: number analyzed (Participants) | 11 | 1
  Leukocytes: <0.65* LLN and >60% Decrease from Baseline | 0 | 0
  Leukocytes:>1.5* ULN and >100% Increase from Baseline: number analyzed (Participants) | 11 | 1
  Leukocytes:>1.5* ULN and >100% Increase from Baseline | 0 | 0
  Basophils/Leukocytes: >4.0* ULN and >300% Increase from Baseline: number analyzed (Participants) | 11 | 1
  Basophils/Leukocytes: >4.0* ULN and >300% Increase from Baseline | 0 | 0
  Eosinophils/Leukocytes: >4.0* ULN and >300% Increase from Baseline: number analyzed (Participants) | 11 | 1
  Eosinophils/Leukocytes: >4.0* ULN and >300% Increase from Baseline | 0 | 0
  Lymphocytes/Leukocytes: <0.25* LLN and >75% Decrease from Baseline: number analyzed (Participants) | 11 | 1
  Lymphocytes/Leukocytes: <0.25* LLN and >75% Decrease from Baseline | 0 | 0
  Lymphocytes/ Leukocytes: >1.5*ULN and >100% Increase from Baseline: number analyzed (Participants) | 11 | 1
  Lymphocytes/ Leukocytes: >1.5*ULN and >100% Increase from Baseline | 0 | 0
  Monocytes/Leukocytes: >4.0* ULN and >300% Increase from Baseline: number analyzed (Participants) | 11 | 1
  Monocytes/Leukocytes: >4.0* ULN and >300% Increase from Baseline | 0 | 0
  Neutrophils/Leukocytes: <0.65*LLN and >75% Decrease from Baseline: number analyzed (Participants) | 11 | 1
  Neutrophils/Leukocytes: <0.65*LLN and >75% Decrease from Baseline | 0 | 0
  Neutrophils/Leukocytes: >1.6*ULN and >100% Increase from Baseline: number analyzed (Participants) | 11 | 1
  Neutrophils/Leukocytes: >1.6*ULN and >100% Increase from Baseline | 0 | 0
  Platelets: <0.65*LLN and >50% Decrease from Baseline: number analyzed (Participants) | 11 | 1
  Platelets: <0.65*LLN and >50% Decrease from Baseline | 0 | 0
  Platelets: >1.5 *ULN and >100% Increase from Baseline: number analyzed (Participants) | 11 | 1
  Platelets: >1.5 *ULN and >100% Increase from Baseline | 1 | 0

19. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Clinical Chemistry Assessments
Description: Criteria for potential clinically significant results were: Aspartate Aminotransferase and Alanine Aminotransferase: >3.0* ULN and >100% increase from baseline (IFB); Bilirubin: >1.5* ULN and >100% IFB; Direct Bilirubin: >2.0* ULN and >150% IFB; Alkaline Phosphatase: 80% decrease from baseline (DFB) and >3.0* ULN and >100% IFB; Urea Nitrogen:100% DFB and >3.0* ULN and >200% IFB; Creatinine >2.0* ULN and >100% IFB; Sodium :10% DFB or >1.1* ULN and >10% IFB; Potassium: 20% DFB or >1.2* ULN and >20% IFB; Chloride: 20% DFB or >1.2*ULN and >20% IFB; Bicarbonate: 40% DFB or >1.3* ULN and >40% IFB; Calcium: 30% DFB or >1.3* ULN and >30% IFB; Albumin: 50% DFB or >1.5* ULN and >50% IFB; Glucose: 40% DFB or >3.0*ULN and >200% IFB.
Time Frame: From first dose of study treatment (Day 1) until TOC (Up to Day 28)
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Aztreonam- Avibactam (ATM- AVI) | Best Available Therapy (BAT)
Number analyzed (Participants) | 12 | 2
Participants
  Aspartate Aminotransferase: >3.0* ULN and >100% Increase from Baseline: number analyzed (Participants) | 11 | 1
  Aspartate Aminotransferase: >3.0* ULN and >100% Increase from Baseline | 1 | 0
  Alanine Aminotransferase: >3.0* ULN and >100% Increase from Baseline: number analyzed (Participants) | 11 | 1
  Alanine Aminotransferase: >3.0* ULN and >100% Increase from Baseline | 0 | 0
  Bilirubin: >1.5* ULN and >100% Increase from Baseline: number analyzed (Participants) | 11 | 1
  Bilirubin: >1.5* ULN and >100% Increase from Baseline | 1 | 0
  Direct Bilirubin: >2.0* ULN and >150% Increase from Baseline: number analyzed (Participants) | 11 | 1
  Direct Bilirubin: >2.0* ULN and >150% Increase from Baseline | 1 | 0
  Alkaline Phosphatase:80% Decrease from Baseline: number analyzed (Participants) | 11 | 1
  Alkaline Phosphatase:80% Decrease from Baseline | 0 | 0
  Alkaline Phosphatase:>3.0* ULN and >100% Increase from Baseline: number analyzed (Participants) | 11 | 1
  Alkaline Phosphatase:>3.0* ULN and >100% Increase from Baseline | 1 | 0
  Urea Nitrogen:100% Decrease from Baseline: number analyzed (Participants) | 11 | 1
  Urea Nitrogen:100% Decrease from Baseline | 0 | 0
  Urea Nitrogen:>3.0* ULN and >200% Increase from Baseline: number analyzed (Participants) | 11 | 1
  Urea Nitrogen:>3.0* ULN and >200% Increase from Baseline | 0 | 0
  Creatinine:>2.0* ULN and >100% Increase from Baseline: number analyzed (Participants) | 11 | 2
  Creatinine:>2.0* ULN and >100% Increase from Baseline | 0 | 0
  Sodium:10% Decrease from Baseline: number analyzed (Participants) | 11 | 1
  Sodium:10% Decrease from Baseline | 0 | 0
  Sodium:>1.1* ULN and >10% Increase from Baseline: number analyzed (Participants) | 11 | 1
  Sodium:>1.1* ULN and >10% Increase from Baseline | 0 | 0
  Potassium:20% Decrease from Baseline: number analyzed (Participants) | 11 | 1
  Potassium:20% Decrease from Baseline | 1 | 0
  Potassium:>1.2* ULN and >20% Increase from Baseline: number analyzed (Participants) | 11 | 1
  Potassium:>1.2* ULN and >20% Increase from Baseline | 0 | 0
  Chloride:20% Decrease from Baseline: number analyzed (Participants) | 11 | 1
  Chloride:20% Decrease from Baseline | 0 | 0
  Chloride:>1.2*ULN and >20% Increase from Baseline: number analyzed (Participants) | 11 | 1
  Chloride:>1.2*ULN and >20% Increase from Baseline | 0 | 0
  Bicarbonate:40% Decrease from Baseline: number analyzed (Participants) | 11 | 1
  Bicarbonate:40% Decrease from Baseline | 0 | 0
  Bicarbonate:>1.3* ULN and >40% Increase from Baseline: number analyzed (Participants) | 11 | 1
  Bicarbonate:>1.3* ULN and >40% Increase from Baseline | 0 | 0
  Calcium:30% Decrease from Baseline: number analyzed (Participants) | 11 | 1
  Calcium:30% Decrease from Baseline | 0 | 0
  Calcium:>1.3* ULN and >30% Increase from Baseline: number analyzed (Participants) | 11 | 1
  Calcium:>1.3* ULN and >30% Increase from Baseline | 0 | 0
  Albumin:50% Decrease from Baseline: number analyzed (Participants) | 11 | 1
  Albumin:50% Decrease from Baseline | 0 | 0
  Albumin:>1.5* ULN and >50% Increase from Baseline: number analyzed (Participants) | 11 | 1
  Albumin:>1.5* ULN and >50% Increase from Baseline | 0 | 0
  Glucose:40% Decrease from Baseline: number analyzed (Participants) | 11 | 1
  Glucose:40% Decrease from Baseline | 0 | 0
  Glucose:>3.0*ULN and >200% Increase from Baseline: number analyzed (Participants) | 11 | 1
  Glucose:>3.0*ULN and >200% Increase from Baseline | 0 | 0

20. Secondary Outcome: Number of Participants With Clinically Significant Abnormalities in Electrocardiogram (ECG)
Description: A standard 12-lead ECG was recorded with the participant in a supine position after at least 10 minutes of rest. The following ECG parameters were recorded: heart rate, PR-interval, QRS-duration, QT-interval, QTc-interval, RR interval. Clinical significance of ECG abnormalities was judged by Investigator.
Time Frame: From first dose of study treatment (Day 1) until TOC (Up to Day 28)
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Aztreonam- Avibactam (ATM- AVI) | Best Available Therapy (BAT)
Number analyzed (Participants) | 12 | 2
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality: From randomization up to late follow-up visit (up to 45 days); SAEs and non-SAEs: From first dose of study drug up to the late follow-up visit (up to maximum of 45 days)
Description: Same event may appear as non-SAE and SAE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study. All-cause mortality is presented for ITT analysis set and non-SAEs and SAEs are presented for safety analysis set.
Arm/Group | Aztreonam- Avibactam (ATM- AVI) | Best Available Therapy (BAT)
All-Cause Mortality (participants affected / at risk) | 2/12 | 1/3
Serious Adverse Events (participants affected / at risk) | 5/12 | 2/2
Other Adverse Events (participants affected / at risk) | 9/12 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aztreonam- Avibactam (ATM- AVI) (N=12) | Best Available Therapy (BAT) (N=2)
Cardiac arrest (Cardiac disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Urinary tract infections (Infections and infestations) | 0 | 1
Bacterial test positive (Investigations) | 1 | 0
Enterococcus test positive (Investigations) | 1 | 0
Neoplasm progession (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aztreonam- Avibactam (ATM- AVI) (N=12) | Best Available Therapy (BAT) (N=2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Ocular hypertension (Eye disorders) | 1 | 0
Frequent bowel movements (Gastrointestinal disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Intervertebral discitis (Infections and infestations) | 1 | 0
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Stoma prolapse (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Catheter culture positive (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Platelet count increased (Investigations) | 1 | 0
Staphylococcus test positive (Investigations) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 0
Device occlusion (Product Issues) | 1 | 0
Intensive care unit delirium (Psychiatric disorders) | 1 | 0
Ureterolithiasis (Renal and urinary disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Skin maceration (Skin and subcutaneous tissue disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Phlebitis (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-05-23): https://cdn.clinicaltrials.gov/large-docs/44/NCT03580044/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-21): https://cdn.clinicaltrials.gov/large-docs/44/NCT03580044/SAP_001.pdf